CLINICAL TRIAL: NCT04908566
Title: Immune Checkpoint Inhibitor PD-1 Antibody Combined With Fluorouracil, Leucovorin, Oxaliplatin and Irinotecan (FOLFIRINOX) Regimen vs. PD-1 Antibody Combined With Oxaliplatin, Tigio (SOX) Regimen During Perioperative Period A Randomized Controlled Phase II Clinical Study for the Treatment of Locally Advanced Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Immune Checkpoint Inhibitor PD-1 Antibody Combined With Chemotherapy in the Perioperative Treatment of Locally Advanced Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJGI-002
Record Dates: First submitted 2021-04-27; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-03

CONDITIONS: Locally Advanced Gastric Adenocarcinoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 antibody combined with FOLFIRINOX regimen (Experimental)
  Interventions: Drug: PD-1 antibody combined with FOLFIRINOX regimen
- PD-1 antibody combined with SOX program (Active Comparator)
  Interventions: Drug: PD-1 antibody combined with SOX program

INTERVENTIONS:
Drug: PD-1 antibody combined with FOLFIRINOX regimen — Give 240 mg of PD-1 antibody before each cycle of chemotherapy, d1; Chemotherapy regimen: irinotecan 150mg/m2, d1; fluorouracil 2400 mg/m², d1-2, continuous pumping for 46 hours; leucovorin 200 mg/m², d1; oxaliplatin 65 mg/m², d1; PD-1 antibody repeats once every 3 weeks; Chemotherapy is repeated every 2 weeks. 4 cycles before surgery. 4 cycles after operation。
  Arms: PD-1 antibody combined with FOLFIRINOX regimen
Drug: PD-1 antibody combined with SOX program — Give 240 mg of PD-1 antibody before each cycle of chemotherapy, d1; Chemotherapy regimen: oxaliplatin 130 mg/m², d1, ticgio 40-60mg bid, d1-14 q3w;Repeat once every 3 weeks.
  2-4 cycles before surgery. The perioperative period was 8 cycles.
  Arms: PD-1 antibody combined with SOX program

SUMMARY:
The FOLFIRINOX regimen has become the standard treatment regimen for advanced colorectal cancer, advanced pancreatic cancer and postoperative adjuvant treatment for pancreatic cancer. With the continuous exploration of Chinese scholars, it has also revised the modified dose suitable for the physical fitness of the Chinese people, which is well tolerated and has a clear efficiency. The drugs in this program are all standard treatment drugs for gastric cancer.

In 2020, JAMA Network Open and JAMA Oncology successively reported the application of FOLFIRINOX in the perioperative period of gastric cancer and the late-stage results of gastric cancer, and they obtained very amazing data respectively.

According to the results of CheckMate-649, the FDA approved Nivolumab combined chemotherapy for first-line treatment of advanced or metastatic gastric cancer, gastroesophageal junction cancer and esophageal adenocarcinoma, regardless of PD-L1 expression. At the same time, this is also the first first-line immunotherapy approved by the FDA for gastric cancer.However, there is no definite conclusion about the preoperative neoadjuvant or perioperative clinical research, so it is necessary to explore the efficacy of PD-1 antibody in the perioperative period.

This study is a single-center, randomized, controlled phase II clinical study. The primary endpoint of the study is the perioperative administration of mFOLFIRINOX regimen combined with PD-1 antibody and D2 radical resection for the treatment of resectable advanced gastric cancer. The deep tumor remission rate (TRG0 and TRG1) , secondary endpoints include pCR rate, 3-year DFS rate, safety, R0 resection rate, D2 radical resection rate, 5-year DFS rate, 5-year OS rate.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age, 75 years of age or less, no gender limitation;
2. Patients with untreated locally advanced resectable adenocarcinoma of the stomach or gastroesophageal junction, with clear pathological diagnosis;
3. According to RECIST 1.1, the efficacy evaluation standard for solid tumors, there were definite measurable and evaluable lesions, with spiral CT lesions ≥1cm；
4. Physical condition score KPS score 80-100 points ；
5. Able to receive systemic chemotherapy;
6. No obvious active bleeding;
7. No history of other malignancies, except cured carcinoma in situ of the cervix, basal carcinoma of the skin or squamous cell carcinoma;
8. Women of childbearing age had negative pregnancy test and had voluntarily taken effective and reliable contraceptive measures during the clinical trial；
9. Sign the informed consent form voluntarily；

Exclusion Criteria:

1. There are distant metastasis or local invasion of adjacent organs；
2. Tumor recurrence;
3. Suffered from or had previously suffered from autoimmune diseases;
4. Past organ transplantation or HIV patients;
5. Allergic to 5-fluorouracil, calcium leucoin, oxaliplatin, or irinotecan, or contraindications to 5-fluorouracil, calcium leucoin, oxaliplatin, or irinotecan exist;
6. Malignant secondary disease dating back to 5 years (exceptions: carcinoma in situ of the cervix, adequately treated basal cell carcinoma of the skin)；
7. Severe non-surgical complications or acute infections；
8. Peripheral polyneuropathy>NCI Grad I；
9. Impaired blood system, liver and kidney function. The evaluation criteria are as follows:

   Blood routine: white blood cells (WBC) <3.0×109/L, neutrophils (ANC) <1.5×109/L, platelets (PLT) <100×109/L, hemoglobin (Hb) <90g/L.

   Liver and kidney function: total bilirubin (TBIL)>1.5 times the upper limit of the normal value; urea nitrogen (BUN)>1.5 times the upper limit of the normal value；Creatinine (Cr)>1.5 times the upper limit of the normal value；Alanine aminotransferase and aspartate aminotransferase (ALT and AST)> 3 times the upper limit of the normal value (without liver metastasis)；Alanine aminotransferase and aspartate aminotransferase (ALT and AST)> 5 times the upper limit of the normal value (for liver metastases)；
10. Subjects with symptomatic brain metastases;
11. Subjects with obvious clinical manifestations of arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency, and severe valvular disease;
12. Subjects with severe bone marrow failure;
13. Psychotic subjects who are difficult to control；
14. Pregnant or lactating subjects;
15. Subjects whom the investigator considers inappropriate to participate in this trial；
16. Include in another clinical trial；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Major pathological response(MPR) | Surgery

SECONDARY OUTCOMES:
Pathological complete response(pCR) | Surgery
Disease-free survival(DFS) rate of 3 years | progression of disease (PD) or death from any cause within 3 years
  Time to relapse or progression of disease (PD) or death from any cause within 3 years from subject screening to first recorded
Disease-free survival(DFS) rate of 5 years | progression of disease (PD) or death from any cause within 5 years
  Time to relapse or progression of disease (PD) or death from any cause within 5 years from subject screening to first recorded

CONTACTS AND LOCATIONS:
Locations (1):
- RuiLiu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol